CLINICAL TRIAL: NCT04177459
Title: Rehabilitation of Adolescents Living With Chronic Fatigue. Health and Quality of Life During the Disease, and How to Remain in School and Spare-time Activities. Testing of a Structured Home-based Rehabilitation Program.
Brief Title: Rehabilitation of Adolescents Living With Chronic Fatigue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Trondheim Kommune (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/1081
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Fatigue Syndrome, Chronic
Keywords: Adolescent; Fatigue; Rehabilitation; Health Promotion; Health-related Quality of Life; Sense of Coherence; Emotions; Mood; Leisure Activities
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health promoting dialogue in addition to treatment as usual (Experimental): Health promoting dialogues in addition to follow-up from primary and secondary health care, and from schools, which is individually customized due to fatigue and other symptoms present.
  Interventions: Behavioral: Health promoting dialogue; Other: standard treatment / treatment as usual
- Treatment as usual (Active Comparator): Follow-up from primary and secondary health care, and from Schools, which is individually customized due to fatigue and other symptoms present..
  Interventions: Other: standard treatment / treatment as usual

INTERVENTIONS:
Behavioral: Health promoting dialogue — Health promoting dialogues based on the salutogenic theory, focusing on resources within and around the individual, and on coping strategies. Seven individual dialogues for each participant, individually adapted due to the fatigue. The intervention is offered in the participants home or at the local hospital, dependent on the participants fatigue and what is preferred.
  Arms: Health promoting dialogue in addition to treatment as usual
Other: standard treatment / treatment as usual — Follow-up from primary and secondary health care, and from schools.

SUMMARY:
Previous studies have shown that health-related quality of life (HRQoL) in adolescents living with chronic fatigue syndrome (CFS/ME) is low if compared with healthy adolescents and adolescents living with other chronic diseases. Effective strategies to improve HRQoL in this group are still lacking. Recently we have observed HRQoL in a group of Norwegian adolescents with CFS/ME (not yet published), which is the background for a new study where we have planned an intervention with health promoting dialogues between patient and nurse, as a strategy to improve HRQoL. In this study we have also opened to include adolescents with other chronic fatigue diagnosis with similar challenges in follow-up as in CFS/ME.

ELIGIBILITY:
Inclusion Criteria:

* chronic fatigue as main symptom (including but not limited to diagnostic codes ICD-10 G93.3 CFS/ME, F48.0 Neurasthenia, R53 Fatigue)
* having undergone an interdisciplinary diagnostic evaluation at The Children's Clinic or at The Fatigue and CFS/ME Outpatient Clinic, St. Olavs hospital during the period 1.8.2019 - 1.4.2020.
* being a pupil or wishing to be a pupil.

Exclusion Criteria:

* not Norwegian speaking
* for any reason unable to read and answer a questionnaire
* for any reason unable to take part in the health promoting dialogues

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | 1 year
  assessed by PedsQL Generic Core scale 4.0

SECONDARY OUTCOMES:
Fatigue Questionnaire | 1 year
  PedsQL Multidimensional Fatigue Questionnaire
Mood and Feelings Questionnaire | 1 year
  Short Mood and Feelings Questionnaire
Self-reported follow-up, School functioning and participation in Leisure activities | 1 year
  Self-report form with yes/no answers regarding follow-up from health care personnel, follow-up from school, school attendance and participation in leisure activities.
EQ-5D-5L | 1 year
  EQ-5D-5L is a 5 dimension and 5 level Questionnaire from the Euro Qol Group (supported by the Euro QolGroup Association and Euro Qol Research Foundation). Health states which is defined by EQ-5D-5L-answers, is assigned a score between 0 and 1 by applying preference weights. In Norway it has been common to use preference weights obtained from a sample of the general population in the UK. Norwegian preference weights will be available in near future. EQ-5D is the name of the instrument and is not an acronym. EQ-5D is the correct term to use in print or verbally.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Selvaag, md phd, Study Director — St. Olavs Hospital; Torstein Baade Rø, md phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Barne og ungdomsklinikken (Children's Clinic), Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
The standard consent form used in this study is developed by the regional ethical committee, and does not include consent to make individual participant data available for other researchers.